CLINICAL TRIAL: NCT01762904
Title: Residual Effect of Chlorhexidine 2% / Isopropyl Alcohol 70% Compared to Triclosan 1% / Isopropyl Alcohol 70%
Brief Title: Residual Effect of Chlorhexidine-alcohol Compared to Triclosan-alcohol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Antisepsia Central (Industry)
Responsible Party: Principal Investigator, Alejandro E. Macias, Principal Investigator, Universidad de Guanajuato
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 385-12
Record Dates: First submitted 2013-01-02; First posted 2013-01-08 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Infectious Diseases
Keywords: Antiseptics; Administration cutaneously; Anti-infecting agents, local
MeSH Terms: conditions — Communicable Diseases | interventions — chlorhexidine gluconate; 2-Propanol; Triclosan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole group of 135 units of measurement (Experimental): The arm is composed of 135 units of measurement, it means, 540 determinations to test 2% chlorhexidine gluconate in 70% isopropyl alcohol and 1% triclosan in 70% isopropyl alcohol and two controls.
  The principal unit of measurement it will be four determinations of bacterial counts in a subject for antiseptics and controls to test each of the application sites, and determination as to each separately sampling for each area for each antiseptic forearm. The same subject may be assessed up to three separate occasions provided only after a minimum period of two weeks between each determination.
  Interventions:
  * Biological: Bacterial culture of the prepared skin's areas with two antiseptics and two controls
  * Other: Preparing skin's areas to be tested with two antiseptics and two controls
  Interventions: Other: Bacterial culture of the prepared skin's areas with two antiseptics and two controls; Other: Preparing skin's areas to be tested with two antiseptics and two controls

INTERVENTIONS:
Other: Bacterial culture of the prepared skin's areas with two antiseptics and two controls — Cultures will be taken with a scrub-cup of 5 cm2 of internal area pressed over the skin previously prepared with the substances, then it added a 3 mL of culture broth (D/E Neutralizing Broth, Difco TM) containing a neutralizing agent as washing solution. The skin will scrub with a sterile rubber policeman for 1 minute and the procedure will be conducted once again. Both aliquots will gather together in a sterile tube, and a sample of 50 microliters will spread in a plate containing a neutralizing agar (D/E neutralizing Agar, Difco TM) and incubate at 35°C for 24 hrs. After incubation, the colonies will be counted.
  Other Names: - Neutralizing agar (D/E neutralizing Agar, Difco TM); - Neutralizing broth (D/E Neutralizing Broth, Difco TM)
Other: Preparing skin's areas to be tested with two antiseptics and two controls — All volunteers will be provided with a neutral soap and shampoo without antiseptics for use during a period of two weeks (phase of stabilization of the skin flora). Two antiseptics (2% chlorhexidine gluconate in 70% isopropyl alcohol and 1% triclosan in 70% isopropyl alcohol) and two controls (Scrub the skin without prior application of any substance and Deionized water redistilled) will be tested as skin antiseptics. The intervention consists of preparing four skin's areas with antiseptics and controls, two in each arm of the volunteer. These ones were approximately 25 cm2 on the forearm for each antiseptic or control. The substances will be applied in an outward circular motion using a sterile swab soaked with the solutions. The solution will remain on the skin for 60 seconds, 3 hours and 24 hours before the bacterial culture will be conducted. For the control where it will be does not apply any substance, the scrub starts immediately.
  Other Names: - 2% chlorhexidine gluconate in 70% isopropyl alcohol; - 1% triclosan in 70% isopropyl alcohol; - Scrub the skin without prior application of any substance; - Deionized water redistilled

SUMMARY:
Currently there are few options for skin antisepsis, commercially antiseptic triclosan is mainly used. To have more options, this study is necessary, where investigators will determine the residual effect of 2% chlorhexidine in 70% isopropyl alcohol and 1% triclosan in 70% isopropyl alcohol and choose the one with the best characteristics for skin antisepsis.

DETAILED DESCRIPTION:
2% chlorhexidine has been used as an antiseptic for invasive procedures, such as the skin preparation for surgery or insertion of intravascular catheters, thereby decreasing the incidence of infections. The preparation of the skin with antiseptics, helps mechanically clean the surface of the skin to be subjected to surgical intervention, removing fat, sweat, dead cells and kill bacteria that are in the skin. It has been shown that 2% chlorhexidine in solution with 70% isopropyl alcohol has greater activity than chlorhexidine in aqueous solution. The constant use of triclosan causes resistance of some microorganisms on some antibiotics.It has been shown that 0.5% of triclosan in 60% alcohol isopropyl chlorhexidine is more effective than alcohol. The aim of the study is to know if 2% chlorhexidine has more residual effect than triclosan 1%, both antiseptic diluted in 70% isopropyl alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* Volunteers who have completed the stabilization phase of skin flora.
* Volunteers who does not taken a shower or bath 24 hours before the test.

Exclusion Criteria:

* Volunteers with a score below 100 Colony Forming Unit per square centimeter (CFU/cm2) of forearm skin surface in the control after the stabilization of the skin flora.
* History of skin allergies or atopy, as well as reactions to alcohol, soaps, iodine, chlorine or latex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guanajuato, León, Guanajuato, Mexico

REFERENCES:
- [Background] Karpanen TJ, Worthington T, Hendry ER, Conway BR, Lambert PA. Antimicrobial efficacy of chlorhexidine digluconate alone and in combination with eucalyptus oil, tea tree oil and thymol against planktonic and biofilm cultures of Staphylococcus epidermidis. J Antimicrob Chemother. 2008 Nov;62(5):1031-6. doi: 10.1093/jac/dkn325. Epub 2008 Aug 13. PMID 18703525
- [Background] McDonnell G, Russell AD. Antiseptics and disinfectants: activity, action, and resistance. Clin Microbiol Rev. 1999 Jan;12(1):147-79. doi: 10.1128/CMR.12.1.147. PMID 9880479
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] Edmiston CE Jr, Seabrook GR, Johnson CP, Paulson DS, Beausoleil CM. Comparative of a new and innovative 2% chlorhexidine gluconate-impregnated cloth with 4% chlorhexidine gluconate as topical antiseptic for preparation of the skin prior to surgery. Am J Infect Control. 2007 Mar;35(2):89-96. doi: 10.1016/j.ajic.2006.06.012. PMID 17327187
- [Background] Swenson BR, Hedrick TL, Metzger R, Bonatti H, Pruett TL, Sawyer RG. Effects of preoperative skin preparation on postoperative wound infection rates: a prospective study of 3 skin preparation protocols. Infect Control Hosp Epidemiol. 2009 Oct;30(10):964-71. doi: 10.1086/605926. PMID 19732018
- [Background] Newman JL, Kaiser NE. Extended activity of healthcare antiseptic products: Manivannan G. Disinfection and decontamination, Principles, applications and related issues. 1st Edition, St. Louis, Missouri, USA. CRC Press Editorial, 2007, Oct: 155-152
- [Background] Boyce JM, Pittet D; Healthcare Infection Control Practices Advisory Committee; HICPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Guideline for Hand Hygiene in Health-Care Settings. Recommendations of the Healthcare Infection Control Practices Advisory Committee and the HIPAC/SHEA/APIC/IDSA Hand Hygiene Task Force. Am J Infect Control. 2002 Dec;30(8):S1-46. doi: 10.1067/mic.2002.130391. PMID 12461507
- [Background] Macias JH, Arreguin V, Munoz JM, Alvarez JA, Mosqueda JL, Macias AE. Chlorhexidine is a better antiseptic than povidone iodine and sodium hypochlorite because of its substantive effect. Am J Infect Control. 2013 Jul;41(7):634-7. doi: 10.1016/j.ajic.2012.10.002. Epub 2013 Feb 4. PMID 23380379
- [Background] Kampf G, Kramer A. Epidemiologic background of hand hygiene and evaluation of the most important agents for scrubs and rubs. Clin Microbiol Rev. 2004 Oct;17(4):863-93, table of contents. doi: 10.1128/CMR.17.4.863-893.2004. PMID 15489352
- [Background] Adams D, Quayum M, Worthington T, Lambert P, Elliott T. Evaluation of a 2% chlorhexidine gluconate in 70% isopropyl alcohol skin disinfectant. J Hosp Infect. 2005 Dec;61(4):287-90. doi: 10.1016/j.jhin.2005.05.015. Epub 2005 Oct 10. PMID 16221509
- [Background] Milstone AM, Passaretti CL, Perl TM. Chlorhexidine: expanding the armamentarium for infection control and prevention. Clin Infect Dis. 2008 Jan 15;46(2):274-81. doi: 10.1086/524736. PMID 18171263
- [Background] Karpanen TJ, Worthington T, Conway BR, Hilton AC, Elliott TS, Lambert PA. Penetration of chlorhexidine into human skin. Antimicrob Agents Chemother. 2008 Oct;52(10):3633-6. doi: 10.1128/AAC.00637-08. Epub 2008 Aug 1. PMID 18676882
- [Background] Small H, Adams D, Casey AL, Crosby CT, Lambert PA, Elliott T. Efficacy of adding 2% (w/v) chlorhexidine gluconate to 70% (v/v) isopropyl alcohol for skin disinfection prior to peripheral venous cannulation. Infect Control Hosp Epidemiol. 2008 Oct;29(10):963-5. doi: 10.1086/590664. PMID 18771405
- [Background] Hibbard JS, Mulberry GK, Brady AR. A clinical study comparing the skin antisepsis and safety of ChloraPrep, 70% isopropyl alcohol, and 2% aqueous chlorhexidine. J Infus Nurs. 2002 Jul-Aug;25(4):244-9. doi: 10.1097/00129804-200207000-00007. PMID 12131506
- [Background] Jones RD, Jampani HB, Newman JL, Lee AS. Triclosan: a review of effectiveness and safety in health care settings. Am J Infect Control. 2000 Apr;28(2):184-96. PMID 10760227
- [Background] D'Arezzo S, Lanini S, Puro V, Ippolito G, Visca P. High-level tolerance to triclosan may play a role in Pseudomonas aeruginosa antibiotic resistance in immunocompromised hosts: evidence from outbreak investigation. BMC Res Notes. 2012 Jan 19;5:43. doi: 10.1186/1756-0500-5-43. PMID 22260715
- [Background] Bedoux G, Roig B, Thomas O, Dupont V, Le Bot B. Occurrence and toxicity of antimicrobial triclosan and by-products in the environment. Environ Sci Pollut Res Int. 2012 May;19(4):1044-65. doi: 10.1007/s11356-011-0632-z. Epub 2011 Nov 5. PMID 22057832
- [Background] McMurry LM, Oethinger M, Levy SB. Triclosan targets lipid synthesis. Nature. 1998 Aug 6;394(6693):531-2. doi: 10.1038/28970. No abstract available. PMID 9707111
- [Background] Levy CW, Roujeinikova A, Sedelnikova S, Baker PJ, Stuitje AR, Slabas AR, Rice DW, Rafferty JB. Molecular basis of triclosan activity. Nature. 1999 Apr 1;398(6726):383-4. doi: 10.1038/18803. No abstract available. PMID 10201369
- [Background] Queckenberg C, Meins J, Wachall B, Doroshyenko O, Tomalik-Scharte D, Bastian B, Abdel-Tawab M, Fuhr U. Absorption, pharmacokinetics, and safety of triclosan after dermal administration. Antimicrob Agents Chemother. 2010 Jan;54(1):570-2. doi: 10.1128/AAC.00615-09. Epub 2009 Oct 12. PMID 19822703
- [Background] Russell AD. Whither triclosan? J Antimicrob Chemother. 2004 May;53(5):693-5. doi: 10.1093/jac/dkh171. Epub 2004 Apr 8. PMID 15073159
- [Background] Bartzokas CA, Gibson MF, Graham R, Pinder DC. A comparison of triclosan and chlorhexidine preparations with 60 per cent isopropyl alcohol for hygienic hand disinfection. J Hosp Infect. 1983 Sep;4(3):245-55. doi: 10.1016/0195-6701(83)90025-7. PMID 6195237
- [Background] White WD. Antibacterial bacteriological swab. Br Med J. 1965; 2:229-230.
- [Background] Hobson DW, Bolsen K. Methods of testing oral and topical antiseptics and antimicrobials. In: Block SS, editor. Disinfection, Sterilization, and Preservation. 5th Ed, Philadelphia [PA]: Lippincott Williams & Wilkins; 2001. p.1329-1359.
- [Background] Alvarez JA, Macias JH, Macias AE, Rodriguez E, Munoz JM, Mosqueda JL, Ponce de Leon S. Povidone-iodine against sodium hypochlorite as skin antiseptics in volunteers. Am J Infect Control. 2010 Dec;38(10):822-5. doi: 10.1016/j.ajic.2010.05.019. PMID 20817318
- [Background] Anderson KF. Antibacterial bacteriological swabs. Br Med J. 1965;2:1123-1124.
- [Background] Williamson P, Kligman AM. A new method for the quantitative investigation of cutaneous bacteria. J Invest Dermatol. 1965 Dec;45(6):498-503. doi: 10.1038/jid.1965.164. No abstract available. PMID 5321315
- [Background] Hanski I, von Hertzen L, Fyhrquist N, Koskinen K, Torppa K, Laatikainen T, Karisola P, Auvinen P, Paulin L, Makela MJ, Vartiainen E, Kosunen TU, Alenius H, Haahtela T. Environmental biodiversity, human microbiota, and allergy are interrelated. Proc Natl Acad Sci U S A. 2012 May 22;109(21):8334-9. doi: 10.1073/pnas.1205624109. Epub 2012 May 7. PMID 22566627
- [Background] Malhotra S, Dharmadasa A, Yentis SM. One vs two applications of chlorhexidine/ethanol for disinfecting the skin: implications for regional anaesthesia. Anaesthesia. 2011 Jul;66(7):574-8. doi: 10.1111/j.1365-2044.2011.06706.x. Epub 2011 May 24. PMID 21609325
- [Background] Tanner J. Methods of skin antisepsis for preventing SSIs. Nurs Times. 2012 Sep 11-17;108(37):20, 22. PMID 23035382
- [Background] Sogawa Y, Kobayashi H, Kajiura T, Nishihara Y. Comparison of residual antimicrobial activity of chlorhexidine-containing antiseptics: An express report. J Healthc Infect 2010;2:32-36.
- [Background] Eiselt D. Presurgical skin preparation with a novel 2% chlorhexidine gluconate cloth reduces rates of surgical site infection in orthopaedic surgical patients. Orthop Nurs. 2009 May-Jun;28(3):141-5. doi: 10.1097/NOR.0b013e3181a469db. PMID 19494763
- [Background] Levy SB. Antibacterial household products: cause for concern. Emerg Infect Dis. 2001;7(3 Suppl):512-5. doi: 10.3201/eid0707.017705. PMID 11485643

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Group of 135 Units of Measurement
Started | 135 (January, 2013)
Completed | 135 (October, 2013)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Whole Group of 135 Units of Measurement
Number analyzed (Participants) | 119
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [20 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Residual Effect of Chlorhexidine 2% / Isopropyl Alcohol 70% Administered Topically
Description: 135 determinations to evaluate residual effect of 2% chlorhexidine in 70% isopropyl alcohol.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. 2% chlorhexidine in 70% isopropyl alcohol was tested. Were prepared the skin area of 25 cm2 randomly selected. The solution remained on the skin for 60s, 3h and 24h, everyone on different days.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: (CFU/cm2)
Groups:
- Whole Group of 135 Units of Measurement: 135 determinations to test 2% chlorhexidine in 70% isopropyl alcohol.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. 2% chlorhexidine in 70% isopropyl alcohol was tested. Were prepared the skin area of 25 cm2 randomly selected. The solution remained on the skin for 60s, 3h and 24h, everyone on different days.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Arm/Group | Whole Group of 135 Units of Measurement
Number analyzed (Participants) | 119
(CFU/cm2)
  0 h | 24 [0 to 120]
  3 h | 48 [12 to 96]
  24 h | 24 [0 to 84]
Statistical Analysis 1: Comparison: Whole Group of 135 Units of Measurement; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

2. Primary Outcome: Evaluate the Residual Effect of Triclosan 1% / Isopropyl Alcohol 70% Administered Topically.
Description: 135 determinations to test 1% triclosan in 70% isopropyl alcohol.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. 1% triclosan in 70% isopropyl alcohol was tested. Were prepared the skin area of 25 cm2 randomly selected. The solution remained on the skin for 60s, 3h and 24h, everyone on different days.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: (CFU/cm2)
Groups:
- Whole Group of 135 Units of Measurement: 135 determinations to test 1% triclosan in 70% isopropyl alcohol.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. 1% triclosan in 70% isopropyl alcohol was tested. Were prepared the skin area of 25 cm2 randomly selected. The solution remained on the skin for 60s, 3h and 24h, everyone on different days.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Arm/Group | Whole Group of 135 Units of Measurement
Number analyzed (Participants) | 119
(CFU/cm2)
  0 h | 48 [0 to 180]
  3 h | 48 [0 to 120]
  24 h | 96 [24 to 192]
Statistical Analysis 1: Comparison: Whole Group of 135 Units of Measurement; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

3. Primary Outcome: Evaluate the Effect on the Skin Flora Application Process of Antiseptics by Sterile Swab
Description: 135 units of measurement to test two controls. Principal unit of measurement: four determinations of bacterial counts in a subject for antiseptics and controls to test each of the application sites.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. Deionized water redistilled (Control 2: Control with scrub) and Scrub the skin without prior application of any substance (Control1: Control without scrub) was tested. Were prepared two skin's areas of 25 cm2 randomly selected. The solution remained on the skin for 60s, 3h and 24h.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Time Frame: 24 hrs
Measure: Median (Inter-Quartile Range); unit: (CFU/cm2)
Groups:
- Whole Group of 135 Units of Measurement: 135 determinations to test two controls: Deionized water redistilled and Scrub the skin without prior application of any substance was tested.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. Deionized water redistilled and Scrub the skin without prior application of any substance was tested.
  Were prepared two skin's areas of 25 cm2 randomly selected. The solution remained on the skin for 60s, 3h and 24h, everyone on different days.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Arm/Group | Whole Group of 135 Units of Measurement
Number analyzed (Participants) | 119
(CFU/cm2)
  Control 1: without scrub 0 h | 480 [288 to 1020]
  Control 2: scrub with Deionized water redisti 0 h | 216 [96 to 348]
  Control 1: without scrub 3 h | 288 [144 to 924]
  Control 2: scrub with Deionized water redisti 3 h | 96 [48 to 372]
  Control 1: without scrub 24 h | 288 [192 to 576]
  Control 2: scrub with Deionized water redisti 24 h | 96 [48 to 384]
Statistical Analysis 1: Comparison: Whole Group of 135 Units of Measurement; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

4. Secondary Outcome: Detect Presence of Allergy or Skin Reaction by the Antiseptic Application
Description: 135 units of measurement to test two antiseptics and two controls. Principal unit of measurement: four determinations of bacterial counts in a subject for antiseptics and controls to test each of the application sites.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. 2% chlorhexidine in 70% isopropyl alcohol and 1% triclosan in 70% isopropyl alcohol, Deionized water redistilled and Scrub the skin without prior application of any substance was tested. We prepared four skin's areas of 25 cm2, two in each forearm. The solution remained on the skin for 60s, 3h and 24h.
  Presence of allergy or any skin reaction at 24 hours after the antiseptic application.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: participants
Groups:
- Whole Group of 135 Units of Measurement: 135 units of measurement to test two antiseptics and two controls. Principal unit of measurement: four determinations of bacterial counts in a subject for antiseptics and controls to test each of the application sites.
  All volunteers was provided with a neutral soap without antiseptics for use of two weeks. 2% chlorhexidine in 70% isopropyl alcohol and 1% triclosan in 70% isopropyl alcohol, Deionized water redistilled and Scrub the skin without prior application of any substance was tested. Were prepared four skin's areas of 25 cm2, two in each forearm. The solution remained on the skin for 60s, 3h and 24h.
  Cultures was taken with a scrub-cup of 5 cm2 pressed over the skin, added a 3 mL of culture broth. The skin was scrub with a sterile rubber policeman for 1 minute and the procedure conducted once again. Both aliquots came together in a sterile tube, a sample of 50 microliters were spread in a plate containing a neutralizing agar and were incubated at 35°C for 24 h.
Arm/Group | Whole Group of 135 Units of Measurement
Number analyzed (Participants) | 119
participants | 0 [0 to 3]

ADVERSE EVENTS:
Arm/Group | Whole Group of 135 Units of Measurement
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No